CLINICAL TRIAL: NCT04592107
Title: The Association of Visceral Adiposity Index With Progression of Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Zelal Adibelli, Assistant Prof. Zelal Adibelli, Uşak University
Other Study IDs: UsakU2
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Obesity, Visceral; Chronic Kidney Diseases; Diabetes Mellitus
Keywords: obesity; chronic kidney disease; diabetes mellitus
MeSH Terms: conditions — Obesity, Abdominal; Renal Insufficiency, Chronic; Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: eGFR — estimated glomerular filtration rate

SUMMARY:
The visceral adiposity index (VAI) has been developed, an indicator for the metabolic function of VAT. Previous studies have confirmed the association between the VAI and CKD prevalence. In this study, we attempted to investigate the association between estimated glomerular filtration rate (eGFR) decline and visceral adiposity.

DETAILED DESCRIPTION:
Data were collected from patients with stage 2-5 CKD aged 18 and 80 years and were not on dialysis. These patients were followed up in the Nephrology Department of the Usak University Research and Training Hospital for at least 1 year between December 2017 and November 2018. This study was approved by the Ethics Committee of Usak University School of Medicine. Of 218 patients with stage 2-5 CKD, only 129 were eligible for the study. The exclusion criteria were as follows: missing data, patients older than 80 years, patients taking cholesterol and lipid lowering drugs and steroids. Demographic data (age, gender, and medical history such as diabetes mellitus and hypertension, medications) were collected from the electronic records of the patients, and physical examinations such as blood pressure measurement after 5 minutes of rest, height, weight, waist circumference (WC) measured at the level midway from the lower rib margin and the iliac crest in the midaxillary line while the patients were standing with their feet 25-30 cm apart were performed. Laboratory samples were collected from the patients, transported to the laboratory, and stored at -80°C until analysis. HbA1c levels were measured using the cation exchange high-performance liquid chromatography system (Variant II Turbo HbA1c analyzer, Bio-Rad Laboratories, Hercules, CA, USA). TG, HDL, uric acid, calcium, phosphorus, bicarbonate, urine protein, and creatinine levels were analyzed with the spectrophotometric method using Architect c8000 automated analyzer and original Abbott kits (Abbott Diagnostics Inc, Park City, IL, USA). Two milliliters of blood was added to ethylenediaminetetraacetic acid (EDTA) (1 mg/ml blood) and mixed thoroughly to perform complete blood count by Mindray BC 6800 (Mindray Bio-Medical Electronics Co., Ltd, Shenzhen, China). Parathyroid hormone (PTH) was analyzed with the electrochemiluminescence method using the ADVIA Centaur analyzer (Siemens Healthcare Diagnostics, Munich, Germany). Serum creatinine levels were measured over a 1-year interval. The eGFR was calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. The stages of CKD were defined according to eGFR as stage 2 mild CKD (eGFR = 89-60 mL/min/1.73m2), stage 3a moderate CKD (eGFR = 45-59 mL/min/1.73m2), stage 3b moderate CKD (eGFR = 30-44 mL/min/1.73m2), stage 4 severe CKD (eGFR = 15-29 mL/min/1.73m2), and stage 5 end-stage CKD (eGFR = <15 mL/min/1.73m2). The eGFR change was calculated as the percentage of change in eGFR in 1 year to baseline eGFR. VAI was calculated using the formula (WC/36.8+(1.89xBMI))x(TG/0.81)x(1.52/HDL) for women and (WC/39.68+(1.88xBMI))x(TG/1.03)x(1.31/HDL) for men. BMI was calculated by dividing weight to square of height.

Data were analyzed with the IBM SPSS 22 statistical program. Descriptive statistics were used to define the main characteristics of the patients. Shapiro-Wilk and Kolmogorov-Smirnoff statistical tests were used to assess the normality of the data. All parameters except parathyroid hormone levels were normally distributed. The correlation between the eGFR difference, VAI values, and other parameters was tested with the Pearson correlation test. The difference between the patients with different CKD stages according to the eGFR change and VAI values were tested by the one-way ANOVA test. The independent samples t-test was used to investigate the difference between patients with and without DM and hypertension according to VAI values and eGFR change. Partial Correlation is used for to investigate the correlation between the two variables, where the effect of other variables is kept constant and controlled for both variables. A p value of less than 0.05 was defined as significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with stage 2-5 CKD
* aged 18 and 80 years
* were not on dialysis
* patients were followed up in the Nephrology Department of the Usak University Research and Training Hospital for at least 1 year between December 2017 and November 2018.

Exclusion Criteria:

* The exclusion criteria were as follows:

missing data, patients older than 80 years, patients taking cholesterol and lipid lowering drugs and/or steroids.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic kidney disease patients who were followed up in the Nephrology Department of the Usak University Research and Training Hospital for at least 1 year between December 2017 and November 2018.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
progression of chronic kidney disease | one year
  increase in eGFR of chronic kidney disease patients in one year

CONTACTS AND LOCATIONS:
Overall Officials: Zelal Adibelli, Principal Investigator — Uşak University
Locations (1):
- Usak University, Uşak, Select One, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kramer H, Luke A, Bidani A, Cao G, Cooper R, McGee D. Obesity and prevalent and incident CKD: the Hypertension Detection and Follow-Up Program. Am J Kidney Dis. 2005 Oct;46(4):587-94. doi: 10.1053/j.ajkd.2005.06.007. PMID 16183412
- [Background] Amato MC, Giordano C. Visceral adiposity index: an indicator of adipose tissue dysfunction. Int J Endocrinol. 2014;2014:730827. doi: 10.1155/2014/730827. Epub 2014 Apr 14. PMID 24829577